CLINICAL TRIAL: NCT04831983
Title: Single-Dose Image-Guided Radiotherapy (IGRT) With Focal Boost to the MRI-defined Macroscopic Tumor Volume for Intermediate Unfavorable and High Risk Prostate Cancer
Brief Title: ABlative Radiotherapy (for) Unfavorable Prostate Tumors
Acronym: ABRUPT
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Stefano Arcangeli, Associate Professor, University of Milano Bicocca
Other Study IDs: ABRUPT
Record Dates: First submitted 2021-03-30; First posted 2021-04-05 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: Unfavorable Prostate Tumors; Stereotactic Body Radiotherapy (SBRT); Volumetric Modulated Arc Therapy (VMAT); Prostate Imaging Reporting and Data System (PI-RADS); Toxicity; Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Published clinical evidence confirms that a single dose of 24 Gy provides unprecedented long-term local control in primary and metastatic prostate cancer with safe toxicity profiles, provided that exposure of surrounding healthy tissues is critically assessed with fulfillment of strict constraints and dose distribution is accomplished using image guidance and tracking tools. In the present trial, intermediate unfavorable and selected high-risk organ-confined prostate cancer patients will undergo Single Dose Radiation Therapy (SDRT) With Focal Boost to the MRI-defined Macroscopic Tumor Volume by means of image-guided volumetric intensity-modulated arc radiotherapy (IGRT-VMAT) and state-of-the-art treatment-planning and quality assurance procedures. Androgen Deprivation Therapy (ADT) type and duration has been set as per standard of care, in accordance with current recommendations and guidelines.

DETAILED DESCRIPTION:
Patients enrolled in this observational prospective trial will be offered image-guided, volumetric modulated radiotherapy (IGRT-VMAT) in a single session (SDRT) of 21 Gy to the whole gland with a simultaneous boost of 24 Gy to the macroscopic PI-RADS driven (4-5) tumour(s). ADT will be prescribed concomitantly, as per standard of care. A real time non-ionizing prostate monitoring will be used to account for intra-fractional errors. If the dose constraints to the normal tissues are at risk, these will be prioritised over the aimed boost dose. The primary endpoint of the trial is the treatment related toxicity measured by the CTCAE v5.0. Secondary endpoints are quality of life in different domains (sexual, rectal , urinary) and biochemical outcome.

Patients will be followed at one month, then every 3 months for the first 12 months and every 6 months thereafter. Quality of Life will be prospectively evaluated through validated tools (ECOG, EPIC, IIEF-5, IPSS, ICIQ-SF) at various timepoints. Percentage or total mean score will be reported according the questionnaires, whether they grade values in a scale or use descriptive statistics. Kaplan-Meier curve analysis of biochemical relapse free survival (b-RFS) at 2 and 5-year bRFS for all patients will be estimated.

ELIGIBILITY:
INCLUSION CRITERIA

* Histologically proven prostate adenocarcinoma;
* Intermediate and High risk disease, as per the NCCN definition;
* N0M0 at staging with standard techniques (Bone Scan and Abdominal CT) or (preferably) Choline or PSMA PET-CT;
* ECOG performance status between 0 and 2;
* Life expectancy of > 5 years, in the opinion of the investigator;
* IPSS score must be ≤ 19 (alpha blockers allowed);

EXCLUSION CRITERIA:

* ≥T3b disease according to the 8th AJCC classification;
* PSA>20 ng/ml at any time point;
* Previous local treatment of the prostate with surgery (radical prostatectomy or cryotherapy);
* Previous radiotherapy to the pelvis;
* Previous invasive malignancy unless disease free for a minimum of 5 years;
* Active Crohn's Disease or Ulcerative Colitis;

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unfavorable Intermediate and Selected High Risk Prostate Cancer (no cT3b and PSA > 20 ng/mL allowed), as per NCCN definition
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v.5.0 | 60 months
  To assess treatment related gastrointestinal (GI) and genitourinary (GU) toxicity for patients who undergo SD RT with focal boost on dominant lesion(s) for intermediate unfavorable and selected high risk organ-confined prostate cancer.

SECONDARY OUTCOMES:
QUALITY OF LIFE (QOL) assessed by Expanded Prostate Cancer Index Composite (EPIC-26) Questionnaire. For each domain minimum symptom score (=0) means best QOL and maximum symptom score (=12) means worst QOL | 60 months
  To measure symptom scores for each QOL domain (urinary incontinence, urinary irritative/obstructive, bowel, sexual) after SDRT by EPIC-26 Questionnaire
Number of participants with erectile dysfunction assessed by International Index of Erectile Function Questionnaire ranging from 5 (worst ) to 25 (best) | 60 months
  To assess erectile function after SDRT using IIEF 5
Number of participants with voiding symptoms assessed by International Prostatic Symptoms Score (IPSS), ranging from 0 (best) to 35 (worst) | 60 months
  To assess voiding symptoms after SDRT using IPSS
Number of participants with urinary incontinence assessed by International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), ranging from 0 (best) to 21 (worst) | 60 months
  To assess urinary continence after SDRT using ICIQ-SF
Number of participants with biochemical relapse assessed by PSA (Phoenix definition) | 60 months
  To assess biochemical outcome after SDRT using serum PSA levels

CONTACTS AND LOCATIONS:
Locations (1):
- Radiation Oncology, ASST Monza (University of Milan Bicocca), Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bodo S, Campagne C, Thin TH, Higginson DS, Vargas HA, Hua G, Fuller JD, Ackerstaff E, Russell J, Zhang Z, Klingler S, Cho H, Kaag MG, Mazaheri Y, Rimner A, Manova-Todorova K, Epel B, Zatcky J, Cleary CR, Rao SS, Yamada Y, Zelefsky MJ, Halpern HJ, Koutcher JA, Cordon-Cardo C, Greco C, Haimovitz-Friedman A, Sala E, Powell SN, Kolesnick R, Fuks Z. Single-dose radiotherapy disables tumor cell homologous recombination via ischemia/reperfusion injury. J Clin Invest. 2019 Feb 1;129(2):786-801. doi: 10.1172/JCI97631. Epub 2019 Jan 14. PMID 30480549
- [Result] Zelefsky MJ, Greco C, Motzer R, Magsanoc JM, Pei X, Lovelock M, Mechalakos J, Zatcky J, Fuks Z, Yamada Y. Tumor control outcomes after hypofractionated and single-dose stereotactic image-guided intensity-modulated radiotherapy for extracranial metastases from renal cell carcinoma. Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):1744-8. doi: 10.1016/j.ijrobp.2011.02.040. Epub 2011 May 17. PMID 21596489
- [Result] Brand DH, Tree AC, Ostler P, van der Voet H, Loblaw A, Chu W, Ford D, Tolan S, Jain S, Martin A, Staffurth J, Camilleri P, Kancherla K, Frew J, Chan A, Dayes IS, Henderson D, Brown S, Cruickshank C, Burnett S, Duffton A, Griffin C, Hinder V, Morrison K, Naismith O, Hall E, van As N; PACE Trial Investigators. Intensity-modulated fractionated radiotherapy versus stereotactic body radiotherapy for prostate cancer (PACE-B): acute toxicity findings from an international, randomised, open-label, phase 3, non-inferiority trial. Lancet Oncol. 2019 Nov;20(11):1531-1543. doi: 10.1016/S1470-2045(19)30569-8. Epub 2019 Sep 17. PMID 31540791
- [Result] Foerster R, Zwahlen DR, Buchali A, Tang H, Schroeder C, Windisch P, Vu E, Akbaba S, Bostel T, Sprave T, Zamboglou C, Zilli T, Stelmes JJ, Telkhade T, Murthy V. Stereotactic Body Radiotherapy for High-Risk Prostate Cancer: A Systematic Review. Cancers (Basel). 2021 Feb 12;13(4):759. doi: 10.3390/cancers13040759. PMID 33673077
- [Result] Jackson WC, Silva J, Hartman HE, Dess RT, Kishan AU, Beeler WH, Gharzai LA, Jaworski EM, Mehra R, Hearn JWD, Morgan TM, Salami SS, Cooperberg MR, Mahal BA, Soni PD, Kaffenberger S, Nguyen PL, Desai N, Feng FY, Zumsteg ZS, Spratt DE. Stereotactic Body Radiation Therapy for Localized Prostate Cancer: A Systematic Review and Meta-Analysis of Over 6,000 Patients Treated On Prospective Studies. Int J Radiat Oncol Biol Phys. 2019 Jul 15;104(4):778-789. doi: 10.1016/j.ijrobp.2019.03.051. Epub 2019 Apr 6. PMID 30959121
- [Result] Lukka HR, Pugh SL, Bruner DW, Bahary JP, Lawton CAF, Efstathiou JA, Kudchadker RJ, Ponsky LE, Seaward SA, Dayes IS, Gopaul DD, Michalski JM, Delouya G, Kaplan ID, Horwitz EM, Roach M 3rd, Pinover WH, Beyer DC, Amanie JO, Sandler HM, Kachnic LA. Patient Reported Outcomes in NRG Oncology RTOG 0938, Evaluating Two Ultrahypofractionated Regimens for Prostate Cancer. Int J Radiat Oncol Biol Phys. 2018 Oct 1;102(2):287-295. doi: 10.1016/j.ijrobp.2018.06.008. Epub 2018 Jun 18. PMID 29913254
- [Result] Morgan SC, Hoffman K, Loblaw DA, Buyyounouski MK, Patton C, Barocas D, Bentzen S, Chang M, Efstathiou J, Greany P, Halvorsen P, Koontz BF, Lawton C, Leyrer CM, Lin D, Ray M, Sandler H. Hypofractionated Radiation Therapy for Localized Prostate Cancer: An ASTRO, ASCO, and AUA Evidence-Based Guideline. J Clin Oncol. 2018 Oct 11;36(34):JCO1801097. doi: 10.1200/JCO.18.01097. Online ahead of print. No abstract available. PMID 30307776
- [Result] Macias VA, Barrera-Mellado I. Ultra-hypofractionated radiation therapy for unfavourable intermediate-risk and high-risk prostate cancer is safe and effective: 5-year outcomes of a phase II trial. BJU Int. 2020 Feb;125(2):215-225. doi: 10.1111/bju.14925. Epub 2019 Nov 8. PMID 31614071
- [Result] Widmark A, Gunnlaugsson A, Beckman L, Thellenberg-Karlsson C, Hoyer M, Lagerlund M, Kindblom J, Ginman C, Johansson B, Bjornlinger K, Seke M, Agrup M, Fransson P, Tavelin B, Norman D, Zackrisson B, Anderson H, Kjellen E, Franzen L, Nilsson P. Ultra-hypofractionated versus conventionally fractionated radiotherapy for prostate cancer: 5-year outcomes of the HYPO-RT-PC randomised, non-inferiority, phase 3 trial. Lancet. 2019 Aug 3;394(10196):385-395. doi: 10.1016/S0140-6736(19)31131-6. Epub 2019 Jun 18. PMID 31227373